CLINICAL TRIAL: NCT01551810
Title: The Phase Ⅲ Clinical Trial Protocol for the Influenza Virus Vaccine (Split Virion, Inactivated)
Brief Title: The Clinical Trial Protocol for the Influenza Virus Vaccine (Split Virion, Inactivated)
Acronym: IVV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Hebei Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMBCAMS-04; 2011L01488 (Other: China state food and drug adminstration)
Record Dates: First submitted 2012-03-08; First posted 2012-03-13 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Influenza
Keywords: Influenza Virus Vaccine (Split Virion, Inactivated); Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; vaxigrip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Influenza Virus Vaccine (Experimental): Influenza Virus Vaccine（no Preservative ) 0.5ml intramuscular injections
  Interventions: Biological: Influenza Virus Vaccine; Biological: Influenza Virus Vaccine(contains Preservative)
- Influenza Virus Vaccine(Preservative) (Experimental): Influenza Virus Vaccine（add Preservative ) 0.5ml intramuscular injections
  Interventions: Biological: Influenza Virus Vaccine; Biological: Influenza Virus Vaccine(contains Preservative)

INTERVENTIONS:
Biological: Influenza Virus Vaccine — Influenza Virus Vaccine 0.5ml intramuscular injections
Biological: Influenza Virus Vaccine(contains Preservative) — Influenza Virus Vaccine(contains Preservative)0.5ml intramuscular injections
  Other Names: Vaxigrip

SUMMARY:
The purpose of this study is to evaluate the safety and the immunogenicity of Influenza Virus Vaccine (Split Virion, Inactivated) that do not contains Preservative .

DETAILED DESCRIPTION:
Influenza Virus Vaccine (Split Virion, Inactivated) that do not contains Preservative. HA contents 15μg/0.5ml per dose includ H1N1、H3N2 and B.

Inactivated Split Influenza Vaccine was manufactured by Sanofi Pasteur HA contents 15μg/0.5ml per dose includ H1N1、H3N2 and B.

This is a randomized, blind phase 3 clinical trial. Total 1200 adults (above ages 36 months ) were selected, randomized to two groups [Influenza Virus Vaccine (Split Virion, Inactivated) and Inactivated Split Influenza Vaccine , each group n=600], adults in each group will be vaccinated with one dose of either Influenza Virus Vaccine (Split Virion, Inactivated) or Sanof IVV respectively.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age above 36 months ;
* Adults, parent(s) or guardians are able to understand and sign informed consent for participation;
* Participants or guardians are able to attend all planned clinical appointment and obey and follow all study instructions;
* Infants no vaccinated with influenza or other preventive biologicals in recent 7 days;
* Axillary temperature ≤37℃.

Exclusion Criteria:

* Have medical record of participants or their family on allergy and egg, convulsion, falling sickness, encephalopathy and psychopathy;
* Low platelet or bleeding disorder do not allow vaccination into the muscle;
* Have damaged or lower immunological function;
* Received blood, plasma or immunoglobulin treatment since birth;
* Have inborn abnormality, develop obstacles or clinical diagnostic serious chronic ( Down Syndrome, diabetes, sickle cell anemia or neural Guillain-Barre Syndrome );
* Have or be doubtful of following diseases: respiratory system diseases, acute infection or active chronic, cardiovascular diseases, liver and kidney diseases, skin diseases, HIV.

Min Age: 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and the immunogenicity of Influenza Virus Vaccine (Split Virion, Inactivated) | six months

CONTACTS AND LOCATIONS:
Overall Officials: Guoyang Liao, Ph. D, Principal Investigator — Institute of Medical Biology, Chinese Academy of Medical Sciences; Yuliang Zhao, MD, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Dingxing Center for Disease Prevention and Control, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Jing-Xia G, Yu-Liang Z, Jin-Feng L, Shu-Zhen L, Guo-Yang L, Qi L. Safety and effectiveness assessment of 2011-2012 seasonal influenza vaccine produced in China: a randomized trial. Postgrad Med. 2017 Nov;129(8):907-914. doi: 10.1080/00325481.2017.1369133. Epub 2017 Sep 5. PMID 28825515